CLINICAL TRIAL: NCT01016782
Title: Multi-Center, Double-Blind, Randomized, Vehicle-Controlled, Parallel Group Study of 0444 Gel
Brief Title: Study of 0444 Gel in the Treatment of Inflammatory Lesions of Rosacea
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Fougera Pharmaceuticals Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 0444
Record Dates: First submitted 2009-11-17; First posted 2009-11-19 (Estimated); Last update posted 2014-07-04 (Estimated); Status verified 2014-07

CONDITIONS: Inflammatory Rosacea
Keywords: Inflammatory Rosacea; Rosacea
MeSH Terms: conditions — Rosacea

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (3):
- Test (Experimental): Test product that contains active pharmaceutical ingredient
  Interventions: Drug: 0444
- Reference (Active Comparator): Reference product that contains active pharmaceutical ingredient
  Interventions: Drug: 0444
- Vehicle (Placebo Comparator): Placebo that contains no active pharmaceutical ingredient
  Interventions: Drug: 0444

INTERVENTIONS:
Drug: 0444 — A thin film of gel will be applied and rubbed into the entire face once daily for a period of 70 days

SUMMARY:
The aim of this trial is to assess the efficacy of Metronidazole Topical Gel 1% in the Treatment of Inflammatory Lesions of Rosacea.

Treatment medication will be administered as follows: A thin film of gel will be applied and rubbed into the entire face once daily for a period of 70 days.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of rosacea
* Good health with the exception of rosacea
* Papsules and pustules minimum and maximum requirements

Exclusion Criteria:

* Subjects who are pregnant, nursing, or planning a pregnancy within the study participation period.
* Subjects who have any systemic or dermatological disorders with the exception of rosacea

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 867 (Actual)
Dates: Start 2008-01; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
Reduction in the number of papules and pustules from Baseline to End of Treatment | 70 Days

SECONDARY OUTCOMES:
Reduction in the Investigator's Global Evaluation, Clear or Almost Clear | 70 Days

CONTACTS AND LOCATIONS:
Overall Officials: Angela C Kaplan, Study Director — Fougera Pharmaceuticals Inc.